CLINICAL TRIAL: NCT02683603
Title: Efficacy and Toxicity of Aerosolised Colistin in Ventilator Associated Pneumonia: A Prospective, Randomized Trial
Brief Title: Effect of Aerosolised Colistin in Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Ahlem Trifi, doctor, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tunis university
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: colistin; aerosol; ventilator associated pneumonia; nephrotoxicity; intravenous
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Colistin; Imipenem; Powders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aerosolised (AS) colistin group (Active Comparator): the intervention was: AS colistin and "imipenem. the drug administered was colimycin (colistin) powder 1 million units (MU) by a flakon (Sanofi Winthrop Industry) at the dosage of 4 million units (MU) for 30 minutes 3 times per day for at least 14 days in addition to IV imipenem 1 g three times per day. Nebulisation was made via an ultrasonic vibrating plates nebulizer (Aeroneb Pro® Aerogen Nektar Corporation, Galway, Ireland). Inhaled colimycin® requires specific settings of the ventilator to limit turbulence inspiratory flow. The adjustment consisted in a volume controlled mode with a Tidal volume <8 ml / kg, respiratory rate at 12 cycles / min, I / E: 1/1 and an end inspiratory break > 20%.
  Interventions: Drug: AS colistin and "imipenem"; Drug: AS colimycin (colistin); Drug: AS colistin and imipenem
- intravenous (IV) colistin goup (Active Comparator): the intervention was: IV colistin and "imipenem. the intravenous (IV) colistin goup received IV colimycin (colistin) as a loading dose of 9 MU during 60 minutes followed by 4.5 million units 2 times per day in addition to IV imipenem 1 g three times per day.
  Interventions: Drug: IV colistin " and "imipenem" .; Drug: IV colimycin (colistin); Drug: IV colistin and imipenem

INTERVENTIONS:
Drug: AS colistin and "imipenem" — colimycin (colistin) powder (1 million units (MU) by flakon) by AS route in addition to imipenem
  Other Names: colimycin (colistin) powder (Sanofi laboratories)
  Arms: aerosolised (AS) colistin group
Drug: IV colistin " and "imipenem" . — colimycin (colistin) powder (1 MU by flakon) by intravenous route in addition to imipenem
  Other Names: colimycin (colistin) powder (Sanofi laboratories)
  Arms: intravenous (IV) colistin goup
Drug: AS colimycin (colistin) — nebulisation of colimycin (colistin) for 30 minutes 3 times per day during at least 14 days. Nebulisation was made via an ultrasonic vibrating plates nebulizer (Aeroneb Pro® Aerogen Nektar Corporation, Galway, Ireland).
  Other Names: colimycin (colistin)
  Arms: aerosolised (AS) colistin group
Drug: IV colimycin (colistin) — intravenous colimycin (colistin) : 9 MU during 60 minutes followed by 4.5 million units 2 times per day
  Other Names: colimycin (colistin) powder by intravenous route
  Arms: intravenous (IV) colistin goup
Drug: AS colistin and imipenem — IV imipenem 1 g three times per day.
  Other Names: imipenem
  Arms: aerosolised (AS) colistin group
Drug: IV colistin and imipenem — IV imipenem 1 g three times per day
  Other Names: imipenem
  Arms: intravenous (IV) colistin goup

SUMMARY:
the management of Ventilator-associated pneumonia (VAP) caused by multidrug-resistant (MDR) gram-negative bacilli (GNB) represent a real therapeutic dilemma in intensive care unit (ICU). Colistin remains an effective agent against MDR GNB. However, because of its side effects, mainly nephrotoxicity, other modalities than the intra venous (IV) route should be tried. Several recent data emphasize the interest of inhaled route. The investigators purpose was to evaluate the effectiveness and systemic toxicity of aerosolized colistin in ventilator associated pneumonia.

DETAILED DESCRIPTION:
prospective, randomized, single-blind study comparing two groups of patients treated with aerosolised (AS) colistin versus colistin intravenously (IV). Included were patients who have mechanical ventilation over 48 hours and that have developed a VAP. A VAP was defined as a CPIS (Clinical Pulmonary Infection Score) >6. Exclusion criteria were septic shock and/or bacteraemia. Included patients were divided into two randomized groups. The 1st received colistin in AS as 4 MU by nebulisation 3 times per 24 h. The 2nd received colistin in IV as a loading dose of 9 MU followed by 4.5MU two times per 24 h. Colistin was given for 14 days or until extubation. Patients were followed for 28 days. Therapeutic efficacy was assessed by a primary outcome: the cure of VAP at day 14 of therapy and defined as resolution of clinical and biological signs of infection that means a CPIS< 6 and bacteriological eradication. Secondary outcomes: duration of mechanical ventilation, ICU stay-length and mortality at day 28. Systemic toxicity was assessed by the occurrence of acute renal failure (ARF) defined as increase of plasma creatinine more than 1.5 times its base value.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients older than 18 years, with mechanical ventilation during more than 48 hours, and who have presented a Ventilator associated Pneumonia (VAP) defined as a CPIS (Clinical Pulmonary Infection Score) of more than six

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cure of VAP | day 14 of therapy
  a CPIS (clinical pulmonary infection score) less than 6 and bacterial eradication

SECONDARY OUTCOMES:
occurrence of acute renal failure | From date of randomization until the time of the cessation of colistin, assessed up 14 days on average
  an acute renal failure was defined as increase of plasma creatinine more than 1.5 times its base value.
duration of mechanical ventilation | From date of randomization until the time of weaning from ventilator, an average of 14 days
length of stay in intensive unit | from randomisation until the time of patient discharge, an average of 28 days

OTHER OUTCOMES:
all cause mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahlem Trifi, Study Chair — Tunis University
Locations (1):
- intensive care unit of the University Hospital Center La Rabta, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
yes of course the data is collected on individual cards which identified demographic, clinical and laboratory data for each patient participating. thereafter these data is entered on Statistical Package for Social Sciences (SPSS) software

REFERENCES:
- [Derived] Abdellatif S, Trifi A, Daly F, Mahjoub K, Nasri R, Ben Lakhal S. Efficacy and toxicity of aerosolised colistin in ventilator-associated pneumonia: a prospective, randomised trial. Ann Intensive Care. 2016 Dec;6(1):26. doi: 10.1186/s13613-016-0127-7. Epub 2016 Mar 31. PMID 27033711